CLINICAL TRIAL: NCT03845582
Title: A Phase 2/3 Multicenter, Randomized, Double-masked, Parallel-group, Placebo-controlled Study to Investigate the Safety, Pharmacokinetics, Tolerability, and Efficacy of ALK-001 in Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: Phase 2/3 Study of ALK-001 in Geographic Atrophy
Acronym: SAGA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alkeus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK001-P3001
Record Dates: First submitted 2019-02-15; First posted 2019-02-19 (Actual); Results first posted 2025-10-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2024-11

CONDITIONS: Geographic Atrophy; Age Related Macular Degeneration; AMD; Atrophy, Geographic
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALK-001 (Experimental): Capsule
  Interventions: Drug: ALK-001 oral capsule
- Placebo (Placebo Comparator): Capsule
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ALK-001 oral capsule — Daily administration for 24 months
  Other Names: C20-D3-Retinyl Acetate; C20 Deuterated vitamin A
  Arms: ALK-001
Drug: Placebo oral capsule — Daily administration for 24 months
  Arms: Placebo

SUMMARY:
This is a double-masked, multicenter, randomized, placebo-controlled clinical trial, evaluating the efficacy and safety of ALK-001 in participants with Geographic Atrophy (GA) secondary to age-related macular degeneration (AMD).

Up to 200 participants will receive ALK-001 while up to 100 participants will receive a placebo.

DETAILED DESCRIPTION:
There is no oral treatment available for Geographic Atrophy secondary to AMD. AMD is characterized by an age-related degeneration of the retina.

The root cause for this degeneration or why some people develop AMD while others do not, is unknown. Over 20 years ago, it was hypothesized that the dimerization of vitamin A may be a significant contributor to the etiology of AMD. The eye indeed uses vitamin A as a cofactor to sense light, and a striking chemical signature of the aging and degenerating retina is the accumulation of vitamin A dimers in the retinal pigment epithelium (RPE) and the underlying Bruch's membrane. In rodent models, high levels of vitamin A dimers correlate with poor retinal health, and a variety of mechanisms have been proposed by which vitamin A dimers may induce retinal toxicity. It has been argued that these mechanisms participate in the development and progression of AMD.

ALK-001, the study drug, is a modified form of vitamin A. When taken once a day as a capsule, it replaces natural vitamin A in the body with one that forms vitamin A dimers more slowly. This study will measure the extent to which treatment with ALK-001 slows the progression of Geographic Atrophy.

ELIGIBILITY:
Major Inclusion Criteria:

- At least one eye with geographic atrophy secondary to dry age-related macular degeneration (AMD)

Major Exclusion Criteria:

- Medical condition, which may interfere with the progression of GA, prevent performance of study procedures, compliance with protocol, or continuous participation in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Alkeus Site, Phoenix, Arizona
  - Alkeus Site, Beverly Hills, California
  - Alkeus Site, Lakewood, Colorado
  - Alkeus Site, Clearwater, Florida
  - Alkeus Site, Fort Myers, Florida
  - Alkeus Site, Gainesville, Florida
  - Alkeus Site, Tampa, Florida
  - Alkeus Site, Winter Haven, Florida
  - Alkeus Site, Bloomington, Illinois
  - Alkeus Site, Lexington, Kentucky
  - Alkeus Site, Chevy Chase, Maryland
  - Alkeus Site, Worcester, Massachusetts
  - Alkeus Site, Grand Rapids, Michigan
  - Alkeus Site, Edina, Minnesota
  - Alkeus Site, Northfield, New Jersey
  - Alkeus Site, Great Neck, New York
  - Alkeus Site, Hauppauge, New York
  - Alkeus Site, Cleveland, Ohio
  - Alkeus Site, Ashland, Oregon
  - Alkeus Site, Houston, Texas
  - Alkeus Site-1, San Antonio, Texas
  - Alkeus Site-2, San Antonio, Texas
  - Alkeus Site, Fairfax, Virginia
  - Alkeus Site, Silverdale, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaufman Y, Ma L, Washington I. Deuterium enrichment of vitamin A at the C20 position slows the formation of detrimental vitamin A dimers in wild-type rodents. J Biol Chem. 2011 Mar 11;286(10):7958-7965. doi: 10.1074/jbc.M110.178640. Epub 2010 Nov 12. PMID 21075840
- [Background] Mihai DM, Jiang H, Blaner WS, Romanov A, Washington I. The retina rapidly incorporates ingested C20-D(3)-vitamin A in a swine model. Mol Vis. 2013 Jul 25;19:1677-83. Print 2013. PMID 23914132
- [Background] Saad L, Washington I. Can Vitamin A be Improved to Prevent Blindness due to Age-Related Macular Degeneration, Stargardt Disease and Other Retinal Dystrophies? Adv Exp Med Biol. 2016;854:355-61. doi: 10.1007/978-3-319-17121-0_47. PMID 26427432
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Target enrollment was 200 participants but ultimately only 198 were enrolled.
Period: Overall Study
Arm/Group | ALK-001 | Placebo
Started | 135 | 63
Completed | 94 | 43
Not Completed | 41 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ALK-001 | Placebo | Total
Number analyzed (Participants) | 135 | 63 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 130 | 60 | 190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 45 | 136
  Male | 44 | 18 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 133 | 59 | 192
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 135 | 63 | 198

OUTCOME MEASURES:

1. Primary Outcome: Growth Rate of GA Lesions, as Assessed by Fundus Autofluorescence (FAF)
Time Frame: Baseline to 24 months
Measure: Least Squares Mean (Standard Error); unit: mm2/year
Arm/Group | ALK-001 | Placebo
Number analyzed (Participants) | 135 | 63
mm2/year | 1.62 (0.081) | 1.87 (0.116)

2. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Baseline to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | ALK-001 | Placebo
Number analyzed (Participants) | 135 | 63
Participants | 97 | 52

3. Secondary Outcome: Changes in Visual Acuity
Description: Changes in LLVA and BCVA
Time Frame: Baseline to 24 months
Measure: Least Squares Mean (Standard Error); unit: letters
Arm/Group | ALK-001 | Placebo
Number analyzed (Participants) | 135 | 63
letters
  LLVA | -3.896 (1.316) | -8.298 (1.835)
  BCVA | -6.862 (1.251) | -10.161 (1.771)

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | ALK-001 | Placebo
All-Cause Mortality (participants affected / at risk) | 5/135 | 1/63
Serious Adverse Events (participants affected / at risk) | 26/135 | 14/63
Other Adverse Events (participants affected / at risk) | 59/135 | 34/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ALK-001 (N=135) | Placebo (N=63)
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 5 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Unresponsive to stimuli (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Corona virus infection (Infections and infestations) | 0 | 3
Infection (Infections and infestations) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peritoneal carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Death (General disorders) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ALK-001 (N=135) | Placebo (N=63)
Blood triglycerides increased (Investigations) | 15 | 5
Blood alkaline phosphatase increased (Investigations) | 10 | 5
Glomerular filtration rate decreased (Investigations) | 6 | 4
Corona virus infection (Infections and infestations) | 7 | 6
Urinary tract infection (Infections and infestations) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3
Fall (Injury, poisoning and procedural complications) | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT03845582/Prot_002.pdf
  • Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT03845582/SAP_003.pdf